CLINICAL TRIAL: NCT04039282
Title: Exploring the Use of myfood24 (an Online Nutritional Assessment Tool) in Clinical Dietetic Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other); British Dietetic Association (Unknown); Dietary Assessment Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STH19780
Record Dates: First submitted 2019-07-26; First posted 2019-07-31 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2019-09

CONDITIONS: Nutritional Disorders; Nutrition Therapy; Food Habits
Keywords: nutrition; dietary recall
MeSH Terms: conditions — Nutrition Disorders; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Participant (Other): Patients will be asked to complete an 3 days worth of an online dietary recall prior to their out patient appointment with the dietitian
  Interventions: Device: myfood24
- Dietitian Participant (Other): The Dietitian will be asked to review the patients completed dietary recalls prior to the patient attending their out patient appointment.
  Interventions: Device: myfood24

INTERVENTIONS:
Device: myfood24 — online website for dietary analysis

SUMMARY:
Dietary assessment is a key component of the dietetic care process. Assessments usually take place within dietetic consultations using methods such as 24-hour recall and paper food diaries. This study will examine the feasibility of using an online dietary assessment tool, myfood24 as an alternative to current dietary assessment practices and explore the barriers and facilitators to its use within dietetic clinical practice. This will be a mixed method study using questionnaires and semi structures interviews with both dietitians and patients. Dietitians, and patients with a range of clinical conditions referred to an NHS Dietetic Service, will be recruited. Patients will be asked to trial the system to record their food intake prior to their dietetic appointment. This data will then be used for the dietary assessment within the consultation. Following this, patients and dietitians will be interviewed about their experiences. Quantitative data will be statistically analysed, and thematic analysis will be used to analyse qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Referred to the STH Dietetic Department
* Willing and able to attend a dietetic out-patient appointment
* Can read and understand English
* Have access to the internet
* Willing to engage in technology as part of their care
* Have or willing to obtain their own email address

Exclusion Criteria:

* Under 18 years
* Unable or unwilling to attend a dietetic out-patient appointment
* Unable to read and understand English
* No access to the internet
* Unwilling to engage in technology as part of their care
* Does not have or unwilling to obtain their own email address

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
System Usability | After patients have used the system. Approximately 4 to 8 weeks after baseline.
  System usability score is generated using system usability scale - a validated questionnaire.

SECONDARY OUTCOMES:
Patient Activation | Baseline and end of intervention. (approximately 3 months from baseline)
  Patient activation score will be generated using Patient Activation Measure (PAM) a validated questionnaire.
Acceptability of using the system as part of dietetic care | The acceptability questionnaire and interviews will be completed at the end of the intervention.(approx 3 months from baseline)
  This will be generated using (I) Acceptability questionnaire for patients using a non-validated questionnaire and (2) Through participant interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No